CLINICAL TRIAL: NCT01896765
Title: Intensive Longterm Prevention Program After Myocardial Infarction in Northwest Germany
Brief Title: Intensive Prevention Program After Myocardial Infarction
Acronym: IPP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Herzzentrum Bremen (Other)
Collaborators: Oldenburger Forschungs- und Entwicklungsinstitut für Informatik (OFFIS). (Unknown); University of Luebeck (Other); Klinikum Oldenburg gGmbH (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: BIHKF-7161
Record Dates: First submitted 2013-07-07; First posted 2013-07-11 (Estimated); Last update posted 2020-06-23 (Actual); Status verified 2020-06

CONDITIONS: Myocardial Infarction; Prevention Harmful Effects
MeSH Terms: conditions — Myocardial Infarction

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Intensive prevention program (Experimental): Standard care with respect to medical and interventional therapy plus intensive prevention program with "study nurse"-coordinated education sessions, regular telephone calls, telephone hotline and telemetric care of cardiovascular risk factors (if patient internet connection available).
  Interventions: Behavioral: Intensive Prevention Program; Other: Standard medical and interventional therapy
- Usual care (Other): Standard care with respect to medical and interventional therapy.
  Interventions: Other: Standard medical and interventional therapy

INTERVENTIONS:
Behavioral: Intensive Prevention Program — "Study nurse"-coordinated education sessions, telephone calls, telephone hotline and telemetric care of cardiovascular risk factors (if patient internet connection available).
  Arms: Intensive prevention program
Other: Standard medical and interventional therapy — Medical and interventional therapy following the standard of care.

SUMMARY:
It is unknown, if a modern prevention program, including intense nurse-coordinated education sessions, regular telephone contacts and a telephone hotline for 12 months, significantly reduces cardiovascular risk factors, clinical events and quality of life in myocardial infarction patients compared to usual care. Furthermore, actually no data on the additional effects and the feasibility of longterm telemetric care of cardiovascular risk factors exist.

The primary hypothesis to be tested is that an intensive longterm prevention program compared to the standard of medical care, will achieve better risk factor control and consecutively less clinical adverse events in patients after myocardial infarctions. The study endpoints will be evaluated after 12 months and during long-term course (after 24 months = one year after termination of the prevention program).

In a substudy the effects of short reinterventions ("Prevention Boosts") during long-term course are tested (IPP Prevention Boost Study). Patients with at least one insufficiently controlled risk factor at 24-months visit are randomly assigned to a short (2-month) reintervention vs. no reintervention. The effects of the reinterventions on risk factor control are evaluated after 36 months.

A further substudy focusing on young patients <= 45 years of age at time of MI (IPP-Y = IPP in the Young) was added after completion of the pilot IPP study. In this study we focus on the prevention program in young MI-patients. A retrospective analysis of individual genetic risk (assessed by genetic risk scores) in the young patients is included in this substudy.

ELIGIBILITY:
Inclusion Criteria:

Hospitalisation due to myocardial infarction (ST-elevation or non-ST-elevation myocardial infarction)

Exclusion Criteria:

i) Hemodynamically significant valvular heart disease (> NYHA class II) or inborn cardiac malformations.

ii) Cardiomyopathy associated with hemodynamic obstruction, pregnancy or myocarditis.

iii) Exercise limitations due to clinical conditions not related to CAD. iv) Any major non-cardiac condition that would adversely effect survival during the duration of the study.

v) Patients unlikely to comply to the study treatment and the follow-up visits. vi) Pregnancy (all pre-menopausal females should have a negative serum pregnancy test).

vii) Inability of cooperation with the protocol, including longterm follow-up. viii) Patient refusal or inability to give informed consent. ix) Refusal of the patient's physician regarding trial participation of the patient.

x) Chronic drug or alcohol abuse.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Actual)
Dates: Start 2013-10; Primary Completion 2020-03 (Actual); Study Completion 2020-05 (Actual)

PRIMARY OUTCOMES:
Prevention score (point score of cardiovascular risk factors) | 24 months
Prevention success | 24 months
  Improvement of one of the risk factors LDL-cholesterol, physical inactivity, smoking without deterioration of another (primary endpoint for IPP-Y = substudy on young MI-patients <= 45 years that was added after completion of the pilot study)

SECONDARY OUTCOMES:
Combined endpoint of clinical adverse events | 24 months
Adherence to prognostic relevant medication after myocardial infarction | 24 months

CONTACTS AND LOCATIONS:
Locations (1):
- Herzzentrum Bremen, Bremen, Germany